CLINICAL TRIAL: NCT00943566
Title: A Multicenter, Open-label, Randomized, Parallel Group Study to Compare the Efficacy and Safety of Sufentanil Transdermal System (TDS) With Sustained-Release Morphine Sulfate in Patients With Chronic Pain Due to Cancer
Brief Title: A Safety and Efficacy Study of Sufentanil Transdermal System in Patients With Chronic Pain Due to Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: funding for project discontinued
Sponsor: Labtec GmbH (Industry)
Responsible Party: Peter Klaffenbach, PhD, Labtec GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STDS0901
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Pain
Keywords: Pain; Cancer; Morphine
MeSH Terms: conditions — Chronic Pain; Pain; Neoplasms | interventions — Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sufentanil Transdermal Delivery System (Experimental): Experimental drug
  Interventions: Drug: Sufentanil
- Control (Active Comparator): Sustained release morphine sulfate
  Interventions: Drug: Sustained Release Morphine Sulfate

INTERVENTIONS:
Drug: Sufentanil — Transdermal Delivery System; Apply up to six 3 cm2 sufentanil TDS patches every 3 days for 12 days of observation. The 12 days of observation begin after a 7 day conversion to sustained release morphine sulfate. If the subject continues on the pharmacokinetic portion of the study, an additional 6 days of intervention will be evaluated (at the same dose as the primary efficacy study).
  Arms: Sufentanil Transdermal Delivery System
Drug: Sustained Release Morphine Sulfate — Sustained Release Morphine Sulfate tablets every 12 hours; up to 400 mg every day for 19 days (7 days of conversion to sustained release morphine sulfate and 12 days of observation)
  Arms: Control

SUMMARY:
The study hypothesis is that the safety and efficacy of sufentanil following transdermal application is comparable to sustained release morphine sulphate tablets in patients with chronic pain due to cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the consumption, in milligrams, of rescue analgesia (normal release morphine sulfate tablets) after the administration of sufentanil TDS or sustained release morphine sulfate.

The secondary efficacy objectives of this study are to evaluate:

* Pharmacokinetic data
* Adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 75 with a diagnosis of cancer;
2. If female, is non-pregnant (negative pregnancy test at Visit 1) and non-lactating;
3. If female, is not of childbearing potential
4. Documented history of moderate to severe chronic cancer pain requiring around-the-clock therapy and are likely to benefit from WHO step III opioid analgesics for the duration of the study;
5. Has been informed of the nature of the study and has provided written informed consent;
6. Is willing, able, and competent to complete the entire study and comply with study instructions

Exclusion Criteria:

1. Patient is a pregnant or lactating female (serum pregnancy test conducted at the Screening Visit);
2. Any ongoing serious adverse events (SAEs) at screening and at baseline;
3. Has scheduled elective surgery or other invasive procedures during the period of study participation;
4. Patients with a known intolerance to opioid analgesics or any excipient of the Investigational Product;
5. Patients with respiratory depression with hypoxia and/or hypercapnia, sever chronic obstructive pulmonary disease, cor pulmonale, severe bronchial asthma, paralytic ileus, (obstructive) sleep apnea syndrome;
6. Evidence of clinically significant cardiovascular, renal, hepatic or psychiatric disease, as determined by medical history, clinical laboratory tests, ECG results, and physical examination, that would place the patient at risk upon exposure to the study medication or that may confound the analysis and/or interpretation of the results;
7. Abnormal aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT), or alkaline phosphatase levels (> 3 times the upper level of normal) or an abnormal total bilirubin level (> 1.5 times the upper level of normal) or creatinine clearance < 50 ml/min (calculated using the Cockcroft-Gault formula);
8. Patients with uncontrolled seizures;
9. Patients with increased intracranial pressure;
10. Patients who are receiving hypnotics or other central nervous system (CNS) depressants that, in the opinion of the investigator, may pose a risk of additional CNS depression with opioid medication;
11. Patients with myxoedema, inadequately controlled hypothyroidism or Addisons disease;
12. History of alcohol and/or drug abuse (or a positive urine drug screen at Visit 1) within one year preceding the Screening Visit;
13. Active skin disease;
14. Patients suffering from diarrhea and/or opioid withdrawal;
15. Known positive Hepatitis B or C or HIV status;
16. Has participated in another clinical study of drugs or devices parallel to or < 1 month before study entry, or previous participation in this study;
17. Is an employee of the investigator or study site with direct involvement in the proposed study or other studies under the direction of that investigator or study site, or is a family member of the employees or the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
The consumption (in mg) of rescue analgesia (normal release morphine sulfate tablets) per day after the administration of either sufentanil TDS or SR morphine sulfate. | 6 days

SECONDARY OUTCOMES:
Adverse events | 18 days
Pharmacokinetic data | 6 days